CLINICAL TRIAL: NCT01262469
Title: PHASE II STUDY Evaluating the Toxicity and Activity of the Combination Lapatinib + Capecitabine in Elderly Patients Aged 70 and Over With Metastatic Breast Cancer Over Expressing HER2
Brief Title: Evaluating Lapatinib + Capecitabine in Patients Aged 70 and Over With HER2 Metastatic Breast Cancer.
Acronym: GERICO09
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GERICO 09/0907; 2009-015981-73 (EudraCT Number)
Record Dates: First submitted 2010-12-16; First posted 2010-12-17 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Metastatic Breast Cancer; 70 Years Old Patients and Over; After One Line of Chemotherapy With Trastuzumab
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lapatinib + Capecitabine (Experimental): lapatinib 1250 mg/day (once daily) Capecitabine 2x850 mg/m2/day, days 1-14 during the first cycle and 2x1000 mg/m2/day, days 1-14, every 21 days for following cycles ( if no unacceptable toxicity is observed).
  Interventions: Drug: lapatinib + capecitabine

INTERVENTIONS:
Drug: lapatinib + capecitabine — For Lapatinib: 5 tablets of 250 mg each, once daily, until disease progression or unacceptable toxicity occurence.
  For Capecitabine: 850 mg/m2 twice a day from day 1 to 14 of cycle 1 and 1000 mg/m2 twice a day from day 1 to 14 of the next cycles.
  Other Names: Tyverb; Xeloda

SUMMARY:
GERICO 09/0907 is a Phase II multicentric trial evaluating the toxicity and activity of the combination of lapatinib and capecitabine in locally advanced or metastatic breast cancer over expressing HER2 for patients aged ≥ 70 who have failed after one line of chemotherapy in combination with trastuzumab.

Due to the minimal participation of older people in clinical trials, there is a lack of data to make evidence-based decisions regarding chemotherapy in this indication.

The study is designed to investigate whether elderly patients with locally advanced or metastatic breast cancer over-expressing HER2 could take advantage of the combination lapatinib and capecitabine in term of clinical benefit, and with no adverse effects and no detrimental impact on functional status (part of geriatric assessment).

The main objective is to assess clinical benefit (defined at 4 months as complete response, partial response or stable disease), safety and preserved geriatric independence (main objective is a "bi-criteria" or composite criteria).

DETAILED DESCRIPTION:
More than half of patients who have breast cancer with Her2-positive tumors treated with trastuzumab as a single agent develop resistance within one year of treatment initiation.

Recent studies on this population of patients show that the use of Capecitabine combined with Lapatinib demonstrates an improvement of TTP without an increase of serious toxic effects.

Our study is designed to investigate whether elderly patients with locally advanced or metastatic breast cancer over-expressing HER2 could take advantage of the combination lapatinib (1250mg/day) and capecitabine (1st cycle day 1 to day 14: 850mg/m2/day x2; next cycles day 1 to day 14: 1000 mg/m2/day x2) in term of clinical benefit, and with no adverse effects and no detrimental impact on functional status (part of geriatric assessment). Treatment will continue until disease progression or unacceptable toxicity occurence.

This is a phase II multicentric trial associated to a pharmacokinetic study which aims to assess the effect of age modifications (absorption, distribution, metabolism and elimination) on the combination Lapatinib-Capecitabine by measuring the Cmin-Cmax of both components in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 70
* Histological confirmed advanced breast cancer (metastatic or locally advanced)
* Tumor over expressing HER2 (HER2 3+ in IHC or IHC 2+ and Fish positive) in sample from the primary and/or secondary tumor
* WHO performance status (EGOG) from 0 to 2
* MMS > 25
* Measurable disease (RECIST criteria)
* Progression of disease after one metastatic line of chemotherapy associated with trastuzumab (must be stopped at least 3 weeks before beginning the trial)
* Adequate hematological function (Hb ≥ 10g/dl, ANC ≥ 1500/mm3, platelets ≥ 100 000/mm3)
* Adequate hepatic function (total bilirubine ≤ 1.5ULN, ASAT and ALAT ≤ 3ULN)
* Adequate renal function (measured or calculated creatinine clearance ≥ 40 ml/min - Cockroft)
* LVEF ≥ 50% (US or isotopic method)
* Absence of treatment by enzymatic inhibitors or inducers or any gastric pH modifying agent/drug within a 7-to-14 day period preceding the first administration of one of the trial's products and within the overall duration of the study (see medication list)
* Patients must be affiliated to a Social Security System
* Patient information and written informed consent form signed

Exclusion Criteria:

* Life expectancy < 3 months
* Prior treatment with capecitabine or lapatinib
* Concomitant radiotherapy except for palliative reason and more than 25% of the BM
* Patients with pre-existing toxicity ≥ grade 2 (excepted alopecia)
* Patients with dysphagia, or inability to swallow the capsules.
* Patient with malabsorption syndrome or disease significantly affecting gastro-intestinal function or with major resection of stomach or proximal bowel that could affect absorption of oral drugs
* Patient already included in another therapeutic trial using an experimental drug within 30 days preceding entry into the study
* Individual deprived of liberty or placed under the authority of a tutor
* Patient with any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-12; Primary Completion 2011-12 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Efficacy assessment | at 4 months
  Benefit is defined as complete response, partial response, or stable disease according to RECIST criteria (vers. 1.1).
  Efficacy criteria is the number of patients meeting this definition. Patients having stopped before this 4-months time point will be considered as non responders without clinical benefit.
Tolerance criteria and impact on functional status | at 4 months
  The criteria is the number of patients for whom a toxicity event (according to the NCI-CTC AE vers.4)and/or an impact on functional status (defined by the 8 items IADL assessment scale) has been observed during the first 4 months of treatment.

SECONDARY OUTCOMES:
Duration of clinical benefit | from treatment start until disease progression
Time to progression | from inclusion to disease progression or death due to breast cancer
Overall response rate | from treatment start until end of treatment
Progression free survival | from inclusion to disease progression or death due to any cause
Overall survival | from inclusion until death due to any cause or last follow-up news (censored data)
Time to treatment failure endpoint | from inclusion to end of treatment
  Treatment stop can be due to toxicity, death, refusal to continue study, or progressive disease.
Determination of toxicity of the combination (NCI-CTC vers.4) | from informed consent signature to one month after last study drug intake
Geriatric Evaluation | At baseline, at uneven cycles, at end of treatment and at follow-up visits (every 6 months)
  Activities of daily Living (ADL)/ Instrumental ADL(IADL), Geriatric depression scale (GDS), Mini Mental States (MMS), comorbidities (CIRGS), G8 (oncodage), Vulnerable Elders Survey (VES13), QLQC30 item 29-30.
Determination of the minimal and maximal concentration of lapatinib and capecitabine | at Day1 Cycle1 and Day1 Cycle3
  The samples time points are the followings:
  T0 : before administration of treatment (lapatinib is administered 1 hour before meal and capecitabine 30 min before meal)
  T1 : time for Cmax (2 hrs post-dose lapatinib and 90 min post-dose of capecitabine)
Number of patients treated with 3 and 6 cycles and % of dose administrated | From treatment start until 6 cycles of treament

CONTACTS AND LOCATIONS:
Overall Officials: Véronique GIRRE, Principal Investigator — CHD Vendée
Locations (20):
- France (20):
  - Centre Paul Papin, Angers
  - Centre Hospitalier de Beauvais, Beauvais
  - Clinique Tivoli, Bordeaux
  - Ch Fleyriat, Bourg-en-Bresse
  - Institut Cancérologie- CENTRE HOSPITALIER BREST, Brest
  - Centre Francois Baclesse, Caen
  - Centre Hospitalier de Lagny-Sur-Marne, Lagny-sur-Marne
  - Centre Oscar Lambret, Lille
  - Institut Paoli Calmettes, Marseille
  - Centre Rene Gauducheau, Nantes
  - Centre Antoine Lacassagne, Nice
  - Centre Hospitalier Orleans La Source, Orléans
  - Institut Curie, Paris
  - Hegp-Hopital Broussais, Paris
  - Polyclinique de Courlancy, Reims
  - Centre Hospitalier de Roanne, Roanne
  - Centre Henri Becquerel, Rouen
  - Centre Rene Huguenin, Saint-Cloud
  - Centre Paul Strauss, Strasbourg
  - Institut Claudius Regaud, Toulouse